CLINICAL TRIAL: NCT05326841
Title: Effect of Cholecalciferol Supplementation on Disease Activity and Quality of Life of Systemic Lupus Erythematosus Patients
Brief Title: Effect of Cholecalciferol Supplementation on Disease Activity and Quality of Life of Systemic Lupus Erythematosus Patients .
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Fiblia, student, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cholecalciferol 5000 IU
Record Dates: First submitted 2022-03-23; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Lupus Erythematosus, Systemic; Cholecalciferol Supplementation; Disease Activity; Quality of Life
Keywords: lupus erythematosus systemic; cholecalciferol supplementation; Mex-SLEDAI score; Lupus QoL
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: There are two groups : cholecalciferol group( intervention group) which get cholecalciferol 5000 iu/day for 12 weeks and saccharum lactis group ( placebo group) which get saccharum lactis for 12 weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is a double blinded randomized controlled trial. Subjects were allocated in each treatment arm using permuted block randomization, with a block size of four and concealed code lists. Investigators, doctors, and subjects were blinded to treatment allocation (double blind).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cholecalciferol group (Experimental): Participants in this arm take a vitamin D3 dose 5000 international units (IU) daily by mouth for a duration of 12 weeks
  Interventions: Drug: Vitamin D3
- placebo group (Placebo Comparator): Participants in this arm take a vitamin D3 placebo daily by mouth for a duration of 12 weeks
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — cholecalciferol tablet, the dose is 5000 international unit /day for 12 weeks
  Other Names: Cholecalciferol

SUMMARY:
Increase in the prevalence and survival rates has led to the assessment of disease activity and quality of life of SLE patients as targets in treatment. Cholecalciferol supplementation was considered as having a role in reducing disease activity and improving quality of life.This research was a double blind, randomized, controlled trial was conducted on female outpatients aged 18-60 years with SLE, consecutively recruited from September to December 2021 at Cipto Mangunkusumo Hospital. Sixty subjects who met the research criteria were randomized and equally assigned into the cholecalciferol and placebo groups. The study outcomes were measured at baseline and after 12 weeks of intervention. we measured he level of vitamin D before and after intervention, the disease activity by MEX-SLEDAI score and the quality of life by Lupus QoL

ELIGIBILITY:
Inclusion Criteria:

* Women subjects aged 18-60 years old with hypovitaminosis D

Exclusion Criteria:

* declining consent to participate, late stage chronic kidney disease (staged 4-5), decompensated liver cirrhosis, consumption of glucocorticoids (equivalent to prednisone 20 mg/day) in the past 30 days, pregnant or lactating, patients with acute infection, hypercalcemic patients, anticonvulsant consumption.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — subjects in this research were female
Enrollment: 60 (Actual)
Dates: Start 2021-10-03 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
level of disease activity of participants at 12 weeks | level of vitamin d was measured at 12 weeks after the intervention
  level of disease activity from the participants at 12 weeks as respons from taking vitamin D and placebo by using Mex-sledai with score from 0 until 34. no activity or remission is 0-1, mild 2-5, moderate 6-9, severe 10-13, very severe more than and equally of 14.
Level of quality of life of participants at 12 weeks | level of quality of life was measured at 12 weeks after intervention
  Level of lupus quality of life from the participants at 12 weeks as respsons from taking vitamin d and placebo by using Lupus QoL with score minimal 0, maximal 100. better quality of life > 75

SECONDARY OUTCOMES:
the level vitamin D of participants at 12 weeks | Level of vitamin D was measured at 12 weeks after intervention
  the level of vitamin D from participants at 12 weeks as respons from taking vitamin D3 and placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Rscm Divisi Alergi Imunologi, Jakarta Pusat, Dki Jakarta, Indonesia